CLINICAL TRIAL: NCT02635594
Title: Effects of Carnipure® Tartrate on Postprandial Endothelial Function and Recovery From Physical Exertion in Healthy People - a Randomized, Double-blind, Placebo-controlled, Two-way Cross-over Study
Brief Title: Effects of Carnipure® Tartrate on Postprandial Endothelial Function and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lonza Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: BTS884/15
Record Dates: First submitted 2015-12-10; First posted 2015-12-21 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Volunteers; Recovery; Endothelial Function
MeSH Terms: interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carnipure® tartrate (Experimental): 1000mg of L-Carnitine provided as 1475mg Carnipure® tartrate
  Interventions: Dietary Supplement: L-Carnitine
- Placebo (Placebo Comparator): 1000mg cellulose + 475mg L-tartaric acid
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-Carnitine — 1000mg of L-Carnitine provided as 1475mg Carnipure® tartrate
  Arms: Carnipure® tartrate
Other: Placebo — 1000mg cellulose + 475mg L-tartaric acid
  Arms: Placebo

SUMMARY:
Investigation of 4 weeks supplementation with Carnipure® tartrate on endothelial function and parameters of recovery after physical exertion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 25 and 45 years
* Body mass index (BMI) between 20 and 30 kg/m²
* Non-smoker
* Physically active 1-2 times per week

Exclusion Criteria:

1. Competitive athlete or performance of high intensity training
2. Vegan
3. Nutrition with high portion of meat (> 3 times meat per week).
4. Injury at the finger
5. History or presence of significant cardiovascular disease or co-morbidities (i.e., diabetes, etc.)
6. Known allergy to ingredients of study preparation
7. Disturbed absorption due to changes in the gastrointestinal tract (e.g., resections, diverticula, blind-loop syndrome)
8. Hypo/ hypertension or taking anti hypo/ hypertension medication
9. Untreated thyroid dysfunction
10. Atherosclerosis or other relevant musculoskeletal diseases/ injuries
11. Anemia (women: Hb <11 g/ dl; men: 12.5 g/ dl)
12. Eating disorder
13. Present or recent use of drugs and dietary supplements that affect the endothelial function, re-covery or lipid status 2 months before or during the study (e.g. L-Carnitine, Arginine, omega3 FA, polyphenol rich supplements (e.g. OPC, cacao, etc) antihypertensive drugs, anti hyperlipidemic drugs, regular intake of protein-shakes etc.)
14. Subjects not willing to abstain from intake of analgesic medication 24 hours prior to and during visit 1b and 3b.
15. Female patients that are pregnant or nursing
16. Night shift worker
17. Donation of blood or similar blood loss within the previous 30 days before screening;
18. Participation in a clinical trial with an investigational product within 30 days before screening
19. Known alcohol abuse or drug abuse
20. Known infection of human immunodeficiency virus (HIV) or hepatitis B or C
21. Known lactose intolerance, dairy protein allergy or allergy to nuts

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
postprandial endothelial function | after 4 weeks supplementation
  postprandial endothelial function assessed after 4 weeks supplementation with verum in comparison to placebo

SECONDARY OUTCOMES:
Maximal strength (Nm) before and after exhaustive exercise | immediately before, 0h, 2h, 24h, 48h,
  Maxiaml strength assessed after 4 weeks supplementation with verum in comparison to placebo at different time points, each (pre exhaustive exercise, immediately after, 2h, 24h and 48h after)
pain before and after exhaustive exercise (VAS) | immediately before, 0h, 2h, 24h, 48h,
  Pain assessed after 4 weeks supplementation with verum in comparison to placebo at different time points, each (pre exhaustive exercise, immediately after, 2h, 24h and 48h after)
Creatin Kinase (CK) before and after exhaustive exercise | immediately before, 0h, 2h, 24h, 48h,
  Assessement of CK after 4 weeks supplementation with verum in comparison to placebo at different time points, each (pre exhaustive exercise, immediately after, 2h, 24h and 48h after)
Myoglobine (Mb) before and after exhaustive exercise | immediately before, 0h, 2h, 24h, 48h,
  Assessement of Mb after 4 weeks supplementation with verum in comparison to placebo at different time points, each (pre exhaustive exercise, immediately after, 2h, 24h and 48h after)
Biomarker for vascular health | after 4 weeks supplementation
  Biomarker for vascular health assessed after 4 weeks supplementation with verum in comparison to placebo

OTHER OUTCOMES:
Adverse Events | after 4 weeks supplementation
  Adverse events assessed after 4 weeks supplementation with verum and placebo
Blood routine parameters | at screening and after 4 weeks supplementation
  Blood routine parameters (differentiated haemogram; blood lipids; glucose; kreatinin) as safety parameters assessed at screening and after 4 weeks supplementation with verum and placebo
Tolerability (questionnaire) | after 4 weeks supplementation
  Tolerability assessed after 4 weeks supplementation with verum in comparison to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, PhD, Principal Investigator — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Baden-Wurttemberg, Germany